CLINICAL TRIAL: NCT04187339
Title: A Phase 1, Randomized, Placebo-controlled, Double-blind, Two-part Study to Evaluate the Safety and Tolerability of NGM395 in Adult Obese Patients (Part 1) and in Adult Patients With Nonalcoholic Fatty Liver Disease (NAFLD) (Part 2).
Brief Title: Study of NGM395 in Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGM395-OB-101
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Obesity; NAFLD
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- NGM395 Dose 1 (Experimental): NGM395 Subcutaneous Injection
  Interventions: Biological: NGM395
- NGM395 Dose 2 (Experimental): NGM395 Subcutaneous Injection
  Interventions: Biological: NGM395
- NGM395 Dose 3 (Experimental): NGM395 Subcutaneous Injection
  Interventions: Biological: NGM395
- NGM395 Dose 4 (Experimental): NGM395 Subcutaneous Injection
  Interventions: Biological: NGM395
- NGM395 Dose 5 (Experimental): NGM395 Subcutaneous Injection
  Interventions: Biological: NGM395
- NGM395 Dose 6 (Experimental): NGM395 Subcutaneous Injection
  Interventions: Biological: NGM395
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NGM395 — NGM395 Dose 1
  Arms: NGM395 Dose 1
Biological: NGM395 — NGM395 Dose 2
  Arms: NGM395 Dose 2
Biological: NGM395 — NGM395 Dose 3
  Arms: NGM395 Dose 3
Biological: NGM395 — NGM395 Dose 4
  Arms: NGM395 Dose 4
Biological: NGM395 — NGM395 Dose 5
  Arms: NGM395 Dose 5
Biological: NGM395 — NGM395 Dose 6
  Arms: NGM395 Dose 6
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Study of NGM395 in adult participants.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

1. Body mass index (BMI) in the range of 27 - 45 kg/m², inclusive, at screening, with maximum body weight of 140 kg.

   Part 2:
2. Liver fat ≥8% as assessed by MRI-PDFF.
3. BMI in the range of 27 - 45 kg/m2, inclusive, with maximum body weight of 140 kg at screening.
4. Waist circumference > 40 inches for males or > 35 inches for females.

Exclusion Criteria:

Part 1:

1. Diagnosed with type 2 diabetes (T2D) and/or the use of metformin, dipeptidyl peptidase-4 (DPP4) inhibitors, sodium/glucose cotransporter 2 (SGLT2) inhibitors, sulfonylurea agents, acarbose, or insulin for T2D within 3 months prior to Screening.
2. Subjects with T2D managed with diet alone with HbA1c level > 6.5% or fasting glucose ≥ 126 mg/dL at Screening.
3. History of bariatric surgery.
4. Fasting triglycerides > 400 mg/dL at Screening.

   Part 2:
5. Diagnosed with type 2 diabetes with a HbA1c >9.5%, on thiazolidinediones, sodium/glucose cotransporter 2 (SGLT2) inhibitors, acarbose, or insulin for T2D within 3 months prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs) | 140 Days
  The number and percent of patients reporting treatment emergent adverse events (TEAEs) by cohort.

SECONDARY OUTCOMES:
Serum Concentration of NGM395 | 140 Days
  NGM395 concentration data by cohort

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals, Inc
Locations (1):
- NGM Clinical Study Site, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No